CLINICAL TRIAL: NCT00702767
Title: Tolerance of Increased Infusion Rates of Intravenous Fat Emulsions in Very Low Birth Weight Infants During the First Week of Life
Brief Title: Tolerance of Increased Infusion Rates of Intravenous Fat Emulsions in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OSF Healthcare System (Other)
Responsible Party: Dr. Kamlesh S. Macwan, Neonatalogist, Children's Hospital of Illinois at OSF-Saint Francis Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-060; NCT00516997 (obsolete NCT alias)
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Low Birth Weight
Keywords: This study was completed in October 2006

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: INTRALIPIDS — INTRAVENOUS FAT EMULSIONS

SUMMARY:
This study was completed in October 2006. No further participates are being recruited.

ELIGIBILITY:
Inclusion Criteria:

* All infants who are Appropriate for Gestational Age at Birth and who have a birthweight between 750-1500 grams will be enrolled in this study.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2005-07; Primary Completion 2006-10 (Actual); Study Completion 2007-04 (Actual)

REFERENCES:
- [Derived] Drenckpohl D, McConnell C, Gaffney S, Niehaus M, Macwan KS. Randomized trial of very low birth weight infants receiving higher rates of infusion of intravenous fat emulsions during the first week of life. Pediatrics. 2008 Oct;122(4):743-51. doi: 10.1542/peds.2007-2282. PMID 18829797